CLINICAL TRIAL: NCT01988714
Title: Cognitive Remediation of Schizophrenia in a Community Mental Health Setting
Acronym: SECT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: R01MH068725 (NIH)
Record Dates: First submitted 2013-11-13; First posted 2013-11-20 (Estimated); Last update posted 2019-04-05 (Actual); Status verified 2019-04

CONDITIONS: Experimental Condition TCT; Controlled Condition CG
Keywords: Targeted cognitive training (TCT) plus evidence-based SE; Computer games (CG) plus evidence-based SE
MeSH Terms: interventions — Thrombin Time

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- (TCT) plus evidence-based SE (Experimental): (TCT) plus evidence-based SE
  Interventions: Other: (CG) plus evidence-based SE
- (CG) plus evidence-based SE (Placebo Comparator): (CG) plus evidence-based SE
  Interventions: Other: (TCT) plus evidence-based SE

INTERVENTIONS:
Other: (TCT) plus evidence-based SE — Targeted cognitive computer training (TCT) plus evidence-based SE in a community setting
  Arms: (CG) plus evidence-based SE
Other: (CG) plus evidence-based SE — (CG) plus evidence-based SE
  Arms: (TCT) plus evidence-based SE

SUMMARY:
The purpose of this study is to investigate the usefulness of neuroscience-guided cognitive training combined with community-based supported employment for people with schizophrenia. The investigators will examine the effectiveness of moving our study of neuroplasticity-based restorative targeted cognitive training out of the laboratory and into the community setting; and the investigators will also investigate its utility in enhancing functional outcome in chronically mentally ill adults who are participating in supported employment.

DETAILED DESCRIPTION:
Neurocognitive functioning will be assessed at baseline (study entry), after cognitive training (6 months), and at 12 month follow-up, using the MATRICS Consensus Cognitive Battery (MCCB). The investigators will assess the following six constructs identified by MATRICS as separable, fundamental dimensions of cognitive impairment in schizophrenia, with a likely sensitivity to intervention [26]: 1) Speed of Processing, 2) Attention/Vigilance, 3) Working Memory, 4) Verbal Learning and Memory, 5) Visual Learning and Memory, and 6) Reasoning and Problem Solving (executive functioning). The investigators will also administer the delayed memory trials of HVLT and BVMT, Trails B, and D-KEFS Color-Word Interference Test [27], and will make one modification to the MCCB in utilizing BACS Tower of London [28] in place of NAB Mazes.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of schizophrenia or schizoaffective disorder(DSM-IV criteria)
* between the ages of 18-65
* English as primary language (learned before age 12)
* no major medical or neurological disorder that precludes participation in the study

Exclusion Criteria:

* We will not exclude subjects with substance abuse or dependence as we wish to investigate the real-world effectiveness of this cognitive remediation approach when combined with SE. As per the clinical policy at Community Services, however, patients will not be permitted to attend the SE program or to participate in the study if they are acutely intoxicated. Subjects who miss 5 consecutive days of participation due to intoxication will be dropped and a replacement subject will be recruited.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2009-09; Primary Completion 2016-09-26 (Actual); Study Completion 2016-09-26 (Actual)

PRIMARY OUTCOMES:
Neurocognition improvement | 24 months
  Schizophrenia subjects who receive 80 hours of targeted cognitive training (TCT) plus evidence-based SE in a community setting will show, compared to baseline, greater improvements in neurocognition at 10 weeks, 20 weeks, 6 months, 12 months, 18 months, and 24 months than subjects who receive 80 hours of computer games (CG) plus SE.

SECONDARY OUTCOMES:
employment | 24 months
  Schizophrenia participants who receive 80 hours of TCT plus SE will have higher rates of employment 12, 18, and 24 months than those who receive 80 hours of CG plus SE.

CONTACTS AND LOCATIONS:
Overall Officials: Sophia Vinogradov, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- vinogradov research lab SFVAMC, San Francisco, California, United States

REFERENCES:
- [Derived] Roberts MT, Lloyd J, Valimaki M, Ho GW, Freemantle M, Bekefi AZ. Video games for people with schizophrenia. Cochrane Database Syst Rev. 2021 Feb 4;2(2):CD012844. doi: 10.1002/14651858.CD012844.pub2. PMID 33539561
- [Derived] Biagianti B, Fisher M, Neilands TB, Loewy R, Vinogradov S. Engagement with the auditory processing system during targeted auditory cognitive training mediates changes in cognitive outcomes in individuals with schizophrenia. Neuropsychology. 2016 Nov;30(8):998-1008. doi: 10.1037/neu0000311. Epub 2016 Sep 12. PMID 27617637